CLINICAL TRIAL: NCT03627637
Title: The Effects of Soy on Brain Vascular Function in Elderly Men and Women
Brief Title: Soy and Brain Vascular Function
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Maastricht University Medical Center (Other)
Collaborators: Alpro Foundation (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Prevention
Other Study IDs: METC183017
Record Dates: First submitted 2018-07-24; First posted 2018-08-13 (Actual); Last update posted 2020-01-18 (Actual); Status verified 2020-01

CONDITIONS: Brain Vascular Function; Cerebral Blood Flow; Glucose Metabolism; Cognitive Performance

STUDY DESIGN:
Intervention Model Description: Participants will receive, in random order, daily 70 g of soy nuts (soy treatment) or no food products (control treatment) for sixteen weeks, separated by a wash-out period of at least 8 weeks.
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental: Soy nuts (Experimental)
  Interventions: Dietary Supplement: Soy nuts
- Control - no soy nuts (No Intervention)

INTERVENTIONS:
Dietary Supplement: Soy nuts — Study volunteers will receive daily 70 g of soy nuts (roasted soybeans containing approximately 100 mg isoflavones). The amount of soy protein provided by the nuts equals the FDA recommended daily intake of 25-30 g.
  Arms: Experimental: Soy nuts

SUMMARY:
Cognitive performance is negatively related to an impaired glucose metabolism, possibly due to impairments in brain vascular function. Supported by the statement from the American Heart and American Stroke Association that healthy plant-based diets, which consist of soy foods, protect against cognitive decline, we now hypothesize that soy-induced changes in glucose metabolism cause beneficial effects on brain vascular function thereby improving cognitive performance. The primary objective of this intervention study is thus to evaluate in elderly men and women the effect of a 16-week soy intervention on cerebral blood flow, as quantified by the non-invasive gold standard magnetic resonance imaging (MRI) perfusion method Arterial Spin Labeling (ASL). Cerebral blood flow is a robust and sensitive physiological marker of brain vascular function. Secondary objectives are to examine effects on glucose metabolism using the oral glucose tolerance test and cognitive performance as assessed with a neurophysiological test battery.

ELIGIBILITY:
Inclusion Criteria:

* Aged between 60-70 years
* BMI between 20-30 kg/m2
* Fasting plasma glucose < 7.0 mmol/L
* Fasting serum total cholesterol < 8.0 mmol/L
* Fasting serum triacylglycerol < 4.5 mmol/L
* Systolic blood pressure < 160 mmHg and diastolic blood pressure < 100 mmHg
* Stable body weight (weight gain or loss < 3 kg in the past three months)
* Willingness to give up being a blood donor from 8 weeks before the start of the study, during the study and for 4 weeks after completion of the study
* No difficult venipuncture as evidenced during the screening visit

Exclusion Criteria:

* Allergy or intolerance to soy
* Current smoker, or smoking cessation < 12 months
* Diabetic patients
* Familial hypercholesterolemia
* Abuse of drugs
* More than 3 alcoholic consumptions per day
* Use of soy products or dietary supplements known to interfere with the main outcomes as judged by the principal investigators
* Use medication to treat blood pressure, lipid or glucose metabolism
* Use of an investigational product within another biomedical intervention trial within the previous 1-month
* Severe medical conditions that might interfere with the study, such as epilepsy, asthma, kidney failure or renal insufficiency, chronic obstructive pulmonary disease, inflammatory bowel diseases, auto inflammatory diseases and rheumatoid arthritis
* Active cardiovascular disease like congestive heart failure or cardiovascular event, such as an acute myocardial infarction or cerebrovascular accident
* Contra-indications for MRI imaging (e.g. pacemaker, surgical clips/material in body, metal splinter in eye, claustrophobia)

Ages: 60 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 23 (Actual)
Dates: Start 2018-08-15 (Actual); Primary Completion 2019-12-31 (Actual); Study Completion 2019-12-31 (Actual)

PRIMARY OUTCOMES:
Brain vascular function | Difference between outcomes at the end of a 16-week soy nut intervention and control period.
  Cerebral blood flow as quantified non-invasively by the MRI perfusion method Arterial Spin Labeling (ASL)

SECONDARY OUTCOMES:
Glucose metabolism | Difference between outcomes at the end of a 16-week soy nut intervention and control period.
  Oral Glucose Tolerance Test (OGTT)
Cognitive performance | Difference between outcomes at the end of a 16-week soy nut intervention and control period.
  Cambridge Neuropsychological Test Automated Battery (CANTAB)

OTHER OUTCOMES:
Other physiological parameters: Peripheral vascular function (1) | Difference between outcomes at the end of a 16-week soy nut intervention and control period.
  Flow-mediated vasodilation (FMD)
Other physiological parameters: Peripheral vascular function (2) | Difference between outcomes at the end of a 16-week soy nut intervention and control period.
  Carotid artery reactivity (CAR)
Other physiological parameters: Peripheral vascular function (3) | Difference between outcomes at the end of a 16-week soy nut intervention and control period.
  Pulse wave analysis (PWA)
Other physiological parameters: Peripheral vascular function (4) | Difference between outcomes at the end of a 16-week soy nut intervention and control period.
  pulse wave velocity (PWV)
Other physiological parameters: Peripheral vascular function (5) | Difference between outcomes at the end of a 16-week soy nut intervention and control period.
  Retinal images
Other physiological parameters: Blood pressure | Difference between outcomes at the end of a 16-week soy nut intervention and control period.
  Office and 24-hour ambulatory blood pressure
Other physiological parameters: Continuous blood glucose | Difference between outcomes at the end of a 16-week soy nut intervention and control period.
  36-hour glycaemic response
Other physiological parameters: Advanced glycation endproducts | Difference between outcomes at the end of a 16-week soy nut intervention and control period.
  Serum protein-bound advanced glycation endproducts (AGEs)
Other physiological parameters: Conventional metabolic risk markers (1) | Difference between outcomes at the end of a 16-week soy nut intervention and control period.
  Lipids and Lipoproteins
Other physiological parameters: Conventional metabolic risk markers (2) | Difference between outcomes at the end of a 16-week soy nut intervention and control period.
  Glucose
Other physiological parameters: Conventional metabolic risk markers (3) | Difference between outcomes at the end of a 16-week soy nut intervention and control period.
  Insulin
Other physiological parameters: Conventional metabolic risk markers (4) | Difference between outcomes at the end of a 16-week soy nut intervention and control period.
  Markers for low-grade systemic inflammation
Other physiological parameters: Conventional metabolic risk markers (5) | Difference between outcomes at the end of a 16-week soy nut intervention and control period.
  Markers for microvascular function
Other physiological parameters: Other parameters (1) | Difference between outcomes at the end of a 16-week soy nut intervention and control period.
  Brain-derived neurotrophic factor (blood)
Other physiological parameters: Other parameters (2) | Difference between outcomes at the end of a 16-week soy nut intervention and control period.
  Cortisol levels (saliva)
Other physiological parameters: Parameters for compliance | Difference between outcomes at the end of a 16-week soy nut intervention and control period.
  Isoflavone levels (urine and blood)
Other perceivable benefits: Quality of Life | Difference between outcomes at the end of a 16-week soy nut intervention and control period.
  The Quality of life (QoL) will be assessed using a 32-item questionnaire
Other perceivable benefits: Sleep characteristics | Difference between outcomes at the end of a 16-week soy nut intervention and control period.
  Sleep characteristics will be assessed using the 10-item Pittsburgh Sleep Quality Index
Other perceivable benefits: Mood | Difference between outcomes at the end of a 16-week soy nut intervention and control period.
  Mood will be tested using the Affect Grid
Other perceivable benefits: Physical fitness (1) | Difference between outcomes at the end of a 16-week soy nut intervention and control period.
  Timed up-and-go test (TUGT)
Other perceivable benefits: Physical fitness (2) | Difference between outcomes at the end of a 16-week soy nut intervention and control period.
  The 6-minute walk test (6 MWT)
Other perceivable benefits: Physical fitness (3) | Difference between outcomes at the end of a 16-week soy nut intervention and control period.
  Handgrip test
Other perceivable benefits: Physical fitness (4) | Difference between outcomes at the end of a 16-week soy nut intervention and control period.
  Muscle strength test

CONTACTS AND LOCATIONS:
Overall Officials: Peter J Joris, PhD, Principal Investigator — Maastricht University Medical Center
Locations (1):
- Maastricht University Medical Center, Maastricht, Limburg, Netherlands

REFERENCES:
- [Derived] Tischmann L, Adam TC, Mensink RP, Joris PJ. Longer-term soy nut consumption improves vascular function and cardiometabolic risk markers in older adults: Results of a randomized, controlled cross-over trial. Clin Nutr. 2022 May;41(5):1052-1058. doi: 10.1016/j.clnu.2022.03.014. Epub 2022 Mar 14. PMID 35395555
- [Derived] Kleinloog JPD, Tischmann L, Mensink RP, Adam TC, Joris PJ. Longer-term soy nut consumption improves cerebral blood flow and psychomotor speed: results of a randomized, controlled crossover trial in older men and women. Am J Clin Nutr. 2021 Dec 1;114(6):2097-2106. doi: 10.1093/ajcn/nqab289. PMID 34510189